CLINICAL TRIAL: NCT02235259
Title: A Phase II, Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of XG-104 Ophthalmic Solutions in the Environment, and During Challenge in the Controlled Adverse Environmental (CAESM ) Model for the Treatment of Dry Eye
Brief Title: Efficacy and Safety of XG-104 for the Treatment of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xigen SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDD-1004-059
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- XG-104 low dose (Experimental)
  Interventions: Drug: XG-104
- XG-104 intermediate dose (Experimental)
  Interventions: Drug: XG-104
- XG-104 high dose (Experimental)
  Interventions: Drug: XG-104
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XG-104 — Comparison of XG-104 (3 concentrations) versus placebo eye drops efficacy
  Arms: XG-104 high dose; XG-104 intermediate dose; XG-104 low dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to assess the safety and efficacy of XG-104 Ophthalmic Solution compared to placebo for the treatment of the signs and symptoms of dry eye after a 4 week Three Times a Day (TID) treatment period

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written informed consent
* Have a subject reported history of dry eye
* Have a history of use or desire to use eye drops

Exclusion Criteria:

* Have any clinically significant eye findings that require therapeutic treatment, and/or in the opinion of the Investigator may interfere with study parameters;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used Restasis® within 30 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 4 (or early termination visit) if of childbearing potential.
* Have a known allergy and/or sensitivity to the study drug or its components
* Have a condition or be in a situation which the Investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;
* Be unable or unwilling to follow instructions, including participation in all study assessments and visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining: in the inferior region change from Pre-CAESM to Post- CAESM, as measured by the Ora CalibraTM Scale | Day 29
Worst Dry Eye Symptom | From D22 to Day 28

SECONDARY OUTCOMES:
Fluorescein Staining using Ora Calibra™ Scale and NEI Scale (all régions) Pre- and Post-CAESM | Day 15
Fluorescein Staining using Ora Calibra™ Scale and NEI Scale (all régions) Pre- and Post-CAESM | Day 29
Lissamine Green Staining using Ora Calibra™ Scale and NEI Scale (all regions) (Pre- and Post-CAESM and change from Pre- to Post-CAESM | Day 15
Lissamine Green Staining using Ora Calibra™ Scale and NEI Scale (all regions) (Pre- and Post-CAESM and change from Pre- to Post-CAESM | Day 29
Tear Film Break-up Time (Pre- and Post-CAESM) | Day 15
Tear Film Break-up Time (Pre- and Post-CAESM) | Day 29
Conjunctival Redness using Ora Calibra™ Scale (Pre- and Post-CAESM) | Day 15
Conjunctival Redness using Ora Calibra™ Scale (Pre- and Post-CAESM) | Day 29
Lid Margin Redness using Ora Calibra scale (Pre- and Post-CAESM) | Day 15
Lid Margin Redness using Ora Calibra scale (Pre- and Post-CAESM) | Day 29
Tear Osmolarity (Post-CAESM) | Day 1
Tear Osmolarity (Post-CAESM) | Day 29
Blink Rate (Pre-CAESM ) using Ora Calibra™ Methodology | Day 15
Blink Rate (Pre-CAESM ) using Ora Calibra™ Methodology | Day 29
Ocular Protection Index (OPI 2.0) (Pre-CAESM ) using Ora Calibra™ Methodology | Day 15
Ocular Protection Index (OPI 2.0) (Pre-CAESM ) using Ora Calibra™ Methodology | Day 29
Unanesthetized Schirmer's Test (Pre-CAESM) | Day 15
Unanesthetized Schirmer's Test (Pre-CAESM) | Day 29
Drop Comfort and Symptom Assessment using Ora Calibra™ Scales | Day 1
Drop Comfort and Symptom Assessment using Ora Calibra™ Scales | Day 15
Ocular Surface Disease Index (OSDI) (Pre-CAESM) | Day 15
Ocular Surface Disease Index (OSDI) (Pre-CAESM) | Day 29
Ocular Discomfort using Ora Calibra™ Scale (Pre and Post-CAESM) | Day 15
Ocular Discomfort using Ora Calibra™ Scale (Pre and Post-CAESM) | Day 29
Ocular Discomfort using Ora Calibra™ Discomfort and 4-Symptom Questionnaire (Pre and Post-CAESM) | Day 15
Ocular Discomfort using Ora Calibra™ Discomfort and 4-Symptom Questionnaire (Pre and Post-CAESM) | Day 29
Ocular Discomfort using Ora Calibra™ Scale (during CAESM exposure) | Day 15
Ocular Discomfort using Ora Calibra™ Scale (during CAESM exposure) | Day 29
Daily diary | up to Day 29

OTHER OUTCOMES:
Visual Acuity (ETDRS) (Pre-CAESM) | Day -7
Visual Acuity (ETDRS) (Pre-CAESM) | Day 1
Visual Acuity (ETDRS) (Pre-CAESM) | Day 15
Visual Acuity (ETDRS) (Pre-CAESM) | Day 29
Slit-Lamp Biomicroscopy (Pre- and Post-CAESM) | Day -7
Slit-Lamp Biomicroscopy (Pre- and Post-CAESM) | Day 1
Slit-Lamp Biomicroscopy (Pre- and Post-CAESM) | Day 15
Slit-Lamp Biomicroscopy (Pre- and Post-CAESM) | Day 29
Adverse event query | up to Day 29
Dilated Fundoscopy Biomicroscopy | Day -7
Dilated Fundoscopy Biomicroscopy | Day 29
Intraocular Pressure | Day -7
Intraocular Pressure | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States